CLINICAL TRIAL: NCT02585258
Title: The Glucocorticoid Low-dose Outcome in RheumatoId Arthritis Study Comparing the Cost-effectiveness and Safety of Additional Low-dose Glucocorticoid in Treatment Strategies for Elderly Patients With Rheumatoid Arthritis
Brief Title: The Glucocorticoid Low-dose Outcome in RheumatoId Arthritis Study
Acronym: Gloria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: European Commission (Other)
Responsible Party: Principal Investigator, Prof. dr. M. Boers, Professor, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VUMC-ARC-GLORIA
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: RheumatoId Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Prednisolone; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisolone (Experimental): prednisolone 5 mg per day
  Interventions: Drug: Prednisolone
- placebo (Placebo Comparator): placebo capsules once per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — 1 capsule containing a tablet of 5 mg prednisolone/ day
  Other Names: glucocorticoid
  Arms: prednisolone
Drug: Placebo — 1 capsule containing a placebo tablet / day
  Other Names: matching placebo
  Arms: placebo

SUMMARY:
Comparing the cost-effectiveness and safety of additional low-dose glucocorticoid in treatment strategies for elderly patients with rheumatoid arthritis:

The Glucocorticoid Low-dose Outcome in RheumatoId Arthritis Study (GLORIA)

DETAILED DESCRIPTION:
Rationale: Rheumatoid arthritis (RA) is a condition with high impact both on the individual and society. In the context of comparing the effectiveness of existing healthcare interventions in the elderly, RA is a condition highly relevant to the community since it has a strongly negative impact on the quality of life of the individual, is particularly frequent in the elderly, and is associated with significant costs. RA management remains challenging: there is an urgent unmet medical and societal need for improved treatment strategies that are effective, safe and affordable. Evidence based information on the glucocorticoid (GC) harm/benefit balance will have a high impact on RA treatment strategies and on treatment strategies for the many other inflammatory disorders for which GCs are considered. The Glucocorticoid Low-dose Outcome in RheumatoId Arthritis Study (GLORIA) is a 5-year project funded by the European Commission under the Horizon 2020 Program, designed to address these needs.

Objective: The primary objectives of the GLORIA project are twofold:

1. To assess the effectiveness, safety and cost-effectiveness of low-dose GC therapy (5 mg/day) compared to placebo given for two years as co-treatment for elderly RA patients (≥ 65 years) in a pragmatic randomized trial;
2. To assess study medication adherence through a medication packaging solution, and test the effectiveness of smart device technology to improve adherence.

Other objectives of the GLORIA project are: to deliver an outcome prediction model for individual patient outcome, to tailor treatment strategies for elderly RA patients with comorbidities; and deliver data to support:

1. better guidelines on RA treatment in the elderly;
2. more accurate information for elderly RA patients, their physicians and researchers;
3. improved strategies for trial design and conduct in the elderly.

Study design: The GLORIA study is a randomized, double-blind, placebo-controlled pragmatic multicenter clinical trial to assess the effectiveness and safety of a daily dose of 5 mg prednisolone or matching placebo in elderly RA patients. Patients will be randomized into two arms: the experimental arm (receiving prednisolone 5 mg/day) or the control arm (receiving placebo). The design emulates the routine care setting: eligibility criteria are very liberal, assessments and procedures are tailored to represent standard of care, and concurrent antirheumatic treatment is allowed next to the trial medication with minimal limitations. Furthermore, all patients will have an adherence monitoring device loaded into the cap of the drug bottle; adherence data will be monitored throughout the trial. In addition, to test the effect of adherence reminders, a substudy (another trial) will be nested in the main GLORIA trial.

Substudy design: The substudy is limited to patients with a smart device (smartphone, tablet, etc) who have completed at least 3 months of the main study on treatment. The experimental arm of the substudy will receive an application loaded onto their smart device that communicates with an adherence monitoring device loaded into the cap of the drug bottle and delivers reminders to improve adherence. The control arm of the substudy will not have this application and reminders. The substudy has a duration of three months.

Study population: Patients of 65 years of age and older with RA according to the 1987 or the 2010 classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR), requiring antirheumatic therapy because of inadequate disease control, as evidenced by a disease activity score of 28 joints calculated with erythrocyte sedimentation rate (DAS28) ≥2.60.

Substudy population: Patients in the main study who have completed at least 3 months on treatment, in possession of and familiar with a smart device.

Intervention: In this two-armed clinical trial, patients will be randomized to either the experimental arm or the control arm. The experimental arm will receive prednisolone 5 mg/day added to existing antirheumatic treatment. The control arm will receive matching placebo added to existing antirheumatic treatment. Treatment duration is two years per patient. Subsequently, study drug is tapered in linear fashion to zero in 6 weeks by inserting increasing numbers of non-treatment days. Patients experiencing a flare at that time can restart open label prednisolone at the discretion of the treating rheumatologist.

Co-interventions: As part of standard of care all patients will receive Calcium 500 mg/Vitamin D3 800 IU. Besides the study medication, almost all treatment is allowed; both treatment for comorbidities, as well as antirheumatic treatment. This includes biologic and nonbiologic disease-modifying antirheumatic drugs (DMARDs), non-steroidal anti-inflammatory drugs (NSAIDs), short term oral or parental GCs for comorbidities and acetaminophen. However, it is advised not to start other antirheumatic therapy (DMARD, biologic) or give intra-articular or intramuscular GC injections, especially not in the first 3 months, but it is allowed if clinically judged as unavoidable. In such cases, preferred administration is at baseline.

Substudy intervention: All patients will have an adherence monitoring device loaded into the cap of the drug bottle that will be equipped with a wireless transmitter, which not only tracks adherence but can also communicate real time with a smart device of the patient (smartphone, tablet, etc.), through special software to remind patients of the time of medication. In the substudy, patients with a smart device will receive an application loaded on their smart device that communicates with the adherence monitoring device loaded into the cap of the drug bottle. The app sends a reminder message to the patient when it's time to take the medication and in case of non-adherence the app also sends an alert message to inform the patient he or she has forgotten to take the medication. Eligible patients will be randomized to either the experimental arm that receive reminders on their smart device, or to the control arm that will not receive reminders, for a period of 3 months.

Main study endpoints:

* To measure benefit, primary endpoints are a) signs and symptoms: the time-averaged mean value (estimated from linear mixed models) of the DAS28; b) damage progression: change from baseline after 2-years in total Sharp/van der Heijde damage score of hands and forefeet radiographs.
* To measure safety, the primary endpoint is the total number of patients experiencing at least one serious adverse event, or one clinical event related to the disease or its therapy.
* Other major outcomes are cost-effectiveness, cost-utility, and medication adherence.

Assessment takes place at varying intervals, and includes seven clinic visits and 3 assessments by telephone.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: GLORIA is a pragmatic trial, with measurements that are almost all part of standard of care, and therefore there are no additional risks associated with these measurements. However, the intervention in this trial is that patients are randomized to either standard of care with low-dose GCs or standard of care without low-dose GCs for a duration of two years. It is known that GCs have strong favorable effects on disease activity, of which patients randomised to the control arm (placebo) cannot benefit. However, side effects of GCs are known as well, and patients in the experimental arm (prednisone 5 mg/day) might suffer from them. Although side effects predominantly occur when GC are used in high doses for long periods of time, elderly are more likely to suffer from adverse effects of the disease and its therapy than younger patients. However, elderly are underrepresented or even excluded from many clinical trials, so it is difficult to estimate their risk: this forms the rationale for the trial. To reduce risks, participants are monitored and patients with a low probability of benefit and patients with a high probability of harm will be excluded from participation to this trial. For the substudy to measure adherence through an innovative application, no additional risks are expected: if the application appears to be successful, patients randomised to the intervention can only benefit from it since it improves their medication adherence; in case the application is not successful, for patients not randomised to the application or for patients without a smart device, no difference is expected with the 'normal' situation, in which patients do not have access to an adherence application.

ELIGIBILITY:
Population (base) RA patients of 65 years of age and older requiring antirheumatic therapy.

Inclusion criteria

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* RA according to the 1987 or the 2010 classification criteria of the American College of Rheumatology (ACR) and the European League Against Rheumatism (EULAR) (Aletaha D et al, Ann Rheum Dis 2010;69:1580);
* inadequate disease control, as evidenced by a disease activity score of 28 joints calculated with erythrocyte sedimentation rate (DAS28) ≥2.60;
* age ≥ 65 years.

Exclusion criteria

A potential subject who meets any of the following criteria will be excluded from participation in this study:

Lower probability of benefit:

* Change, stop or start of antirheumatic treatment in the last month prior to eligibility assessment, including methotrexate, sulfasalazine, hydroxychloroquine, leflunomide, azathioprine, intramuscular and oral gold, cyclosporine, biologic agents including anti-tumor necrosis factor (TNF), anakinra, abatacept, rituximab, tocilizumab (temporary exclusion);
* Treatment with systemic GC: oral or parenteral GC with a cumulative prednisolone equivalent dose of 200 mg or higher in the last 3 months;
* Treatment with any GC (oral, intra-articular, intravenous or intramuscular) in the last 30 days (temporary exclusion);
* Note: as this is a pragmatic trial, patients who require start of (other) antirheumatic treatment at baseline or during the trial can still be eligible (see 7.1).

Higher probability of harm:

* Exposure to investigational therapy in the last three months;
* Current participation in another clinical trial;
* Major surgery, donation or loss of approximately 500 ml blood within 4 weeks prior to the screening visit (temporary exclusion)
* Absolute contraindication to low-dose prednisolone, as determined by the treating physician, such as: uncontrolled chronic infections, diabetes mellitus, hypertension, osteoporosis. When these conditions are under control (e.g. with antiosteoporosis drugs, antihypertensive drugs) these patients can enter;
* Absolute contraindication to Calcium and/or Vitamin D supplement as determined by the treating physician, such as: hyperparathyroidism (when insufficiently treated);
* Uncontrolled comorbid conditions, short life span, etc. as determined by the treating physician.

Difficulty to measure harm/benefit:

* Absolute indication to start with oral or intravenous GC, according to the treating physician;
* Inability to comply with medical instructions or inability to assess major outcomes at 6-monthly visits, in the assessment of the treating physician.

Subjects/patients not capable or willing to provide informed consent.

Substudy

Additional exclusion criteria for subjects participating in the substudy to measure the effect of a reminder via smart device on adherence:

Inability/difficulty to measure benefit:

* Not in the possession of a smart device;
* Premature discontinuation of study medication within or at 3 months of the main trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 451 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Boers, Prof. dr., Principal Investigator — Amsterdam UMC, location VUmc
Locations (28):
- Germany (3):
  - Charite, Berlin
  - Facharztpraxis, Magdeburg
  - Knappschaftsklinikum Saar, Püttlingen
- University of Debrecen, Debrecen, Hungary
- University of Genova, Genova, Italy
- Netherlands (15):
  - Noordwest Ziekenhuis, Alkmaar
  - Meander, Amersfoort
  - VUmc, Amsterdam
  - Gelre, Apeldoorn
  - Groene Hart Ziekenhuis, Gouda
  - UMCG, Groningen
  - MCL, Leeuwarden
  - LUMC, Leiden
  - MC Zuiderzee, Lelystad
  - MUMC, Maastricht
  - Maasstad, Rotterdam
  - Antonius Ziekenhuis, Sneek
  - HAGA, The Hague
  - UMC Utrecht, Utrecht
  - VieCurie MC, Venlo
- Portugal (5):
  - CHU Coimbra, Coimbra
  - Hospital de Egas Moniz, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Instituto Portugues de Reumatologia, Lisbon
  - Hospital de Ponte Lima, Ponte de Lima
- Romania (2):
  - Carol Davila University of Medicine and Pharmacy, Bucharest
  - Carol Davila, Bucharest
- NURCH, Bratislava, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
(meta) data will be shared after signing a data sharing agreement, at reasonable cost
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: expected active from 2022
Access Criteria: scientific use

REFERENCES:
- [Background] Palmowski Y, Buttgereit T, Dejaco C, Bijlsma JW, Matteson EL, Voshaar M, Boers M, Buttgereit F. "Official View" on Glucocorticoids in Rheumatoid Arthritis: A Systematic Review of International Guidelines and Consensus Statements. Arthritis Care Res (Hoboken). 2017 Aug;69(8):1134-1141. doi: 10.1002/acr.23185. Epub 2017 Jul 10. PMID 28029750
- [Background] Palmowski Y, Buttgereit F, Boers M. Reply. Arthritis Care Res (Hoboken). 2019 Apr;71(4):577-578. doi: 10.1002/acr.23452. No abstract available. PMID 29073333
- [Background] Hartman L, Rasch LA, Klausch T, Bijlsma HWJ, Christensen R, Smulders YM, Ralston SH, Buttgereit F, Cutolo M, Da Silva JAP, Opris D, Rovensky J, Szamosi S, Middelink LM, Lems WF, Boers M. Harm, benefit and costs associated with low-dose glucocorticoids added to the treatment strategies for rheumatoid arthritis in elderly patients (GLORIA trial): study protocol for a randomised controlled trial. Trials. 2018 Jan 25;19(1):67. doi: 10.1186/s13063-017-2396-3. PMID 29370811
- [Background] Hartman L, Lems WF, Boers M. Outcome measures for adherence data from a medication event monitoring system: A literature review. J Clin Pharm Ther. 2019 Feb;44(1):1-5. doi: 10.1111/jcpt.12757. Epub 2018 Sep 1. PMID 30171815
- [Background] Hartman L, Cutolo M, Bos R, Opris-Belinski D, Kok MR, Griep-Wentink HJRM, Klaasen R, Allaart CF, Bruyn GAW, Raterman HG, Voshaar MJH, Gomes N, Pinto RMA, Klausch LT, Lems WF, Boers M. Medication adherence in older people with rheumatoid arthritis is lower according to electronic monitoring than according to pill count. Rheumatology (Oxford). 2021 Nov 3;60(11):5239-5246. doi: 10.1093/rheumatology/keab207. PMID 33682887
- [Background] Palmowski A, Nielsen SM, Buttgereit T, Palmowski Y, Boers M, Christensen R, Buttgereit F. Association Between Participant Retention and the Proportion of Included Elderly People in Rheumatology Trials: Results From a Series of Exploratory Meta-Regression Analyses. Arthritis Care Res (Hoboken). 2020 Oct;72(10):1490-1496. doi: 10.1002/acr.24051. PMID 31421022
- [Background] Palmowski A, Buttgereit T, Palmowski Y, Nielsen SM, Boers M, Christensen R, Buttgereit F. Applicability of trials in rheumatoid arthritis and osteoarthritis: A systematic review and meta-analysis of trial populations showing adequate proportion of women, but underrepresentation of elderly people. Semin Arthritis Rheum. 2019 Jun;48(6):983-989. doi: 10.1016/j.semarthrit.2018.10.017. Epub 2018 Nov 2. PMID 30466715
- [Background] Palmowski A, Nielsen SM, Buttgereit T, Palmowski Y, Boers M, Christensen R, Buttgereit F. Glucocorticoid-trials in rheumatoid arthritis mostly study representative real-world patients: A systematic review and meta-analysis. Semin Arthritis Rheum. 2020 Dec;50(6):1400-1405. doi: 10.1016/j.semarthrit.2020.02.016. Epub 2020 Mar 2. PMID 32222381
- [Background] Forsat ND, Palmowski A, Palmowski Y, Boers M, Buttgereit F. Recruitment and Retention of Older People in Clinical Research: A Systematic Literature Review. J Am Geriatr Soc. 2020 Dec;68(12):2955-2963. doi: 10.1111/jgs.16875. Epub 2020 Oct 19. PMID 33075140
- [Background] Buttgereit T, Palmowski A, Forsat N, Boers M, Witham MD, Rodondi N, Moutzouri E, Navidad AJQ, Van't Hof AWJ, van der Worp B, Coll-Planas L, Voshaar M, de Wit M, da Silva J, Stegemann S, Bijlsma JW, Koeller M, Mooijaart S, Kearney PM, Buttgereit F. Barriers and potential solutions in the recruitment and retention of older patients in clinical trials-lessons learned from six large multicentre randomized controlled trials. Age Ageing. 2021 Nov 10;50(6):1988-1996. doi: 10.1093/ageing/afab147. PMID 34324628
- [Background] Santiago T, Voshaar M, de Wit M, Carvalho PD, Buttgereit F, Cutolo M, Paolino S, Castelar Pinheiro GR, Boers M, Da Silva JAP. Patients' and rheumatologists' perspectives on the efficacy and safety of low-dose glucocorticoids in rheumatoid arthritis-an international survey within the GLORIA study. Rheumatology (Oxford). 2021 Jul 1;60(7):3334-3342. doi: 10.1093/rheumatology/keaa785. PMID 33394036
- [Background] van der Heijde DM, van Leeuwen MA, van Riel PL, van de Putte LB. Radiographic progression on radiographs of hands and feet during the first 3 years of rheumatoid arthritis measured according to Sharp's method (van der Heijde modification). J Rheumatol. 1995 Sep;22(9):1792-6. PMID 8523365
- [Result] Hartman L, Bos R, Buttgereit F, Guler-Yuksel M, Ionescu R, Kok MR, Lems WF, Micaelo M, Opris-Belinski D, Pusztai A, Santos E, Da Silva J, Szekanecz Z, Zeiner K, Zhang D, Boers M. Remarkable international variability in reasons for ineligibility and non-participation in the GLORIA trial. Scand J Rheumatol. 2019 Jul;48(4):340-341. doi: 10.1080/03009742.2018.1559880. Epub 2019 May 27. No abstract available. PMID 31132016
- [Result] Boers M, Hartman L, Opris-Belinski D, Bos R, Kok MR, Da Silva JA, Griep EN, Klaasen R, Allaart CF, Baudoin P, Raterman HG, Szekanecz Z, Buttgereit F, Masaryk P, Klausch LT, Paolino S, Schilder AM, Lems WF, Cutolo M; GLORIA Trial consortium. Low dose, add-on prednisolone in patients with rheumatoid arthritis aged 65+: the pragmatic randomised, double-blind placebo-controlled GLORIA trial. Ann Rheum Dis. 2022 Jul;81(7):925-936. doi: 10.1136/annrheumdis-2021-221957. Epub 2022 May 31. PMID 35641125
- [Result] Hartman L, da Silva JAP, Buttgereit F, Cutolo M, Opris-Belinski D, Szekanecz Z, Masaryk P, Voshaar MJH, Heymans MW, Lems WF, van der Heijde DMFM, Boers M. Development of prediction models to select older RA patients with comorbidities for treatment with chronic low-dose glucocorticoids. Rheumatology (Oxford). 2023 May 2;62(5):1824-1833. doi: 10.1093/rheumatology/keac547. PMID 36165675
- [Result] Hartman L, El Alili M, Cutolo M, Opris D, Da Silva J, Szekanecz Z, Buttgereit F, Masaryk P, Bos R, Kok MR, Paolino S, Coupe V, Lems WF, Boers M; GLORIA consortium. Cost-effectiveness and cost-utility of add-on, low-dose prednisolone in patients with rheumatoid arthritis aged 65+: The pragmatic, multicenter, placebo-controlled GLORIA trial. Semin Arthritis Rheum. 2022 Dec;57:152109. doi: 10.1016/j.semarthrit.2022.152109. Epub 2022 Oct 21. PMID 36335684
- [Derived] Palmowski A, Nielsen SM, Boyadzhieva Z, Schneider A, Pankow A, Hartman L, Da Silva JAP, Kirwan J, Wassenberg S, Dejaco C, Christensen R, Boers M, Buttgereit F. Safety and efficacy associated with long-term low-dose glucocorticoids in rheumatoid arthritis: a systematic review and meta-analysis. Rheumatology (Oxford). 2023 Aug 1;62(8):2652-2660. doi: 10.1093/rheumatology/kead088. PMID 36810945
- See also: description of DAS28 score instrument — https://www.das-score.nl/en/

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisolone: prednisolone 5 mg per day
  Prednisolone: capsules 5 mg / day
- Placebo: placebo capsules once per day
  Placebo: capsules 1 / day
Period: Overall Study
Arm/Group | Prednisolone | Placebo
Started | 226 | 225
Started Study Meds: Safety Population | 224 | 225
Returned for Follow up: Modified Intention-to-treat (ITT) Population | 221 | 223
Completed | 141 | 137
Not Completed | 85 | 88
Not completed — Adverse Event | 28 | 29
Not completed — Death | 3 | 2
Not completed — Lack of Efficacy | 7 | 9
Not completed — includes covid-related access problems | 42 | 46
Not completed — Lost to Follow-up | 5 | 2

BASELINE CHARACTERISTICS:
Population: safety population: excludes 2 patients who did not start study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Placebo | Total
Number analyzed (Participants) | 224 | 225 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 224 | 225 | 449
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.5 (5.3) | 72.6 (5.4) | 72.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 160 | 156 | 316
  Male | 64 | 69 | 133
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 138 | 145 | 283
  Romania | 27 | 29 | 56
  Italy | 32 | 28 | 60
  Europe | 27 | 23 | 50
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.2 (4.5) | 27.2 (4.4) | 27.2 (4.4)
disease duration [Mean (Standard Deviation); unit: years] | 10.8 (10.4) | 10.2 (10.2) | 10.6 (10.3)
DAS28 (Disease activity scale-28 joints) [Mean (Standard Deviation); unit: units on a scale] — DAS28 is an index that calculates a score based on 4 measures:
  painful joint count (28 joints), swollen joint count (28 joints), patient global assessment (0-10), and erythrocyte sedimentation rate. The range is from 0-8, with higher scores indicating more disease activity.
  see: link in reference list.
  units on a scale | 4.43 (1.04) | 4.60 (1.05) | 4.51 (1.05)
Sharp-van der Heijde damage score [Mean (Standard Deviation); unit: units on a scale] — Sharp van der Heijde joint damage score is a score based on assessment of joint space narrowing and extent of erosions on a semi-quantitative scale, in selected joints of hands and forefeet. Theoretical range is from 0-448. A higher score means more damage.
  See reference list. Population: not all patients had available radiographs for scoring
  units on a scale
    number analyzed (Participants) | 200 | 206 | 406
    (all) | 20.0 (34.6) | 17.2 (33.4) | 18.6 (34.0)

OUTCOME MEASURES:

1. Primary Outcome: Signs and Symptoms: Mean DAS28 Post Baseline
Description: mean of the DAS28 (disease activity score-28 joints) post baseline. Range 0-8, higher scores mean more disease activity. See link in reference list.
Time Frame: 0,3,6,12,18,24 months
Population: modified Intention-to-treat includes all patients who took study medication and attended at least one follow up visit
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 221 | 223
score on a scale
  3 months | 3.26 (0.06) | 3.62 (0.07)
  6 months | 3.06 (0.07) | 3.42 (0.07)
  12 months | 2.89 (0.07) | 3.25 (0.07)
  18 months | 3.02 (0.07) | 3.89 (0.07)
  24 months | 2.97 (0.07) | 3.33 (0.07)
Statistical Analysis 1: Comparison: Prednisolone vs Placebo; mixed model reports the effect of treatment, adjusted for stratification factors; Test type: Superiority; p < 0.0001, Mixed Models Analysis — one-sided; mean difference over 2-years = -0.37, 95% CI 1-sided [upper limit -0.23] — placebo is reference. Negative difference is beneficial, means lower disease activity in prednisolone group

2. Primary Outcome: The Total Number of Patients Experiencing at Least One Adverse Event (AE) of Special Interest (AESI)
Description: AESI: (a serious adverse event [SAE], or an AE on a prespecified list of clinically relevant AEs commonly associated with the disease and glucocorticoid use
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 224 | 225
Participants | 134 | 111
Statistical Analysis 1: Comparison: Prednisolone vs Placebo; mixed model reports the effect of treatment, adjusted for stratification factors; Test type: Superiority; p = 0.02, GEE — one-sided; Risk Ratio (RR) = 1.24, 95% CI 1-sided [lower limit 1.04] — prednisolone/placebo

3. Secondary Outcome: Joint Damage Progression
Description: 2-year change in total Sharp/van der Heijde damage score of hands and forefeet radiographs. Range of damage score: 0-448.
  score at 24 months minus score at baseline: positive result means increasing/worsening of damage.
Time Frame: 0, 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prednisolone | Placebo
Number analyzed (Participants) | 221 | 223
score on a scale | 0.3 (1.0) | 1.9 (6.4)
Statistical Analysis 1: Comparison: Prednisolone vs Placebo; mixed model reports the effect of treatment, adjusted for stratification factors; Test type: Superiority; p = 0.003, Regression, Linear — one-sided; mean differences over 2 years = -1.67, 95% CI 1-sided [upper limit -0.68] — placebo is reference. Negative difference means less damage progression in prednisolone group

ADVERSE EVENTS:
Time Frame: 2 years
Description: At every visit, adjudication of adverse events of special interest (AESI). More details, especially on non-SAE AESI ('other AESI') are reported in the main trial publication (see reference list).
  Specifically for ClinicalTrials.gov, so outside the statistical analysis and reporting plan, we report:
  * SAE per specific term,
  * all non-serious AE reported >5%. This table includes both AESI and non-AESI.
Arm/Group | Prednisolone | Placebo
All-Cause Mortality (participants affected / at risk) | 3/224 | 2/225
Serious Adverse Events (participants affected / at risk) | 55/224 | 46/225
Other Adverse Events (participants affected / at risk) | 169/224 | 164/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=224) | Placebo (N=225)
myocardial infarction (Cardiac disorders) | 3 (4) | 1 (1)
myocardial ischemia (Cardiac disorders) | 1 (1) | 1 (1)
atrial fibrillation/flutter (Cardiac disorders) | 0 (0) | 3 (3)
AV block (Cardiac disorders) | 0 (0) | 1 (1)
cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
cataract (Eye disorders) | 0 (0) | 1 (2)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 3 (3) | 0 (0)
enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
chesst discomfort/pain (General disorders) | 1 (1) | 1 (1)
malaise (General disorders) | 0 (0) | 1 (1)
pyrexia (General disorders) | 1 (1) | 1 (1)
abcess limb (Infections and infestations) | 1 (1) | 0 (0)
appendicitis (Infections and infestations) | 0 (0) | 1 (1)
bursitis infective (Infections and infestations) | 1 (1) | 1 (1)
covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
erysipelas (Infections and infestations) | 0 (0) | 1 (1)
fungal infection (Infections and infestations) | 1 (1) | 0 (0) — oropharyngeal
gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
infectious pleural effusion (Infections and infestations) | 1 (1) | 0 (0)
parainfluenzae infection (Infections and infestations) | 1 (1) | 0 (0)
gastroenteritis, parasitic (Infections and infestations) | 0 (0) | 1 (1)
sepsis (Infections and infestations) | 2 (2) | 1 (1)
septic shock (Infections and infestations) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 7 (8) | 2 (2)
pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
urinary tract infection (Infections and infestations) | 2 (2) | 2 (4)
epidydimitis (Infections and infestations) | 1 (1) | 0 (0)
Postoperative abscess Hematoma infection (Infections and infestations) | 1 (1) | 0 (0)
peritonitis (Infections and infestations) | 0 (0) | 1 (1)
contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — chest
spine fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
pelvic fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — supraspinatus
prostate specific antigen increased (Investigations) | 0 (0) | 1 (1)
weight decrease (Investigations) | 1 (1) | 0 (0)
decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — pseudoseptic
intravertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 3 (3)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
basal cell carinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
epenymoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
gastrointestinal stromal tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
pancreas carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
urothelium transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
carotid atherosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
complex regional pain syndrome (Nervous system disorders) | 0 (0) | 1 (1)
facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 1 (1) | 1 (1)
neuralgia, intercostal (Nervous system disorders) | 1 (1) | 0 (0)
radicular syndrome (Nervous system disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 0 (0) | 2 (2)
transient ischemic attack (Nervous system disorders) | 0 (0) | 2 (2)
intracranial hemorrhage, traumatic (Nervous system disorders) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 2 (2) | 0 (0)
dementia, neuropsychiatric symptoms (Nervous system disorders) | 1 (1) | 0 (0)
urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
cough, productive (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
total hip replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
prostatectomy, transurethral (Surgical and medical procedures) | 0 (0) | 1 (1)
circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=224) | Placebo (N=225)
all nonserious events (General disorders) | 169 (989) | 164 (732) — total. placed under general disorders because system requires an organ system specification
bronchitis, nasopharyngitis, respiratory tract infection (Infections and infestations) | 40 (53) | 36 (50) — combination of 3 terms
urinary tract infection, cystitis (Infections and infestations) | 29 (52) | 16 (30) — combination of terms
influenza, influenza-like illness (Nervous system disorders) | 24 (26) | 22 (25) — combination of terms
pneumonia (Infections and infestations) | 12 (17) | 11 (14)
hypertension (Vascular disorders) | 17 (17) | 14 (14)
headache (Nervous system disorders) | 18 (19) | 7 (7)
cough (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 10 (11)

LIMITATIONS AND CAVEATS:
Initially slow recruitment, initiatives to enhance recruitment and retention hampered or prohibited by strict and varying ethical guidelines across countries.

The covid-19 pandemic compromised collection of important endpoint data. The pragmatic design caused confounding by treatment changes, most likely reducing the difference in benefit between the groups.

Post-hoc specification of adverse event frequencies done outside of statistical analysis plan.

See reference list (trial results).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT02585258/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-02): https://cdn.clinicaltrials.gov/large-docs/58/NCT02585258/SAP_001.pdf